CLINICAL TRIAL: NCT06854640
Title: First in Patient, Dose Escalation, Open Label Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Intravenous Infusion of BAY 3389934 to Patients With Sepsis Induced Coagulopathy
Brief Title: A Study to Learn About How Safe BAY 3389934 is, Its Suitable Dose, and How it Affects the Participants With Sepsis Induced Coagulopathy
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Patient safety concern based on difficulty for investigator to assess coagulation status of patient. Reference is made to the Unexpected Event Notification and associated Safety Report.
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 22265; 2024-515635-30-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2025-02-28; First posted 2025-03-03 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Sepsis; Coagulopathy
Keywords: DIC; Disseminated intravascular coagulation; Sepsis induced coagulopathy
MeSH Terms: conditions — Sepsis; Hemostatic Disorders; Disseminated Intravascular Coagulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dose group 1 of BAY3389934 (Experimental): Subjects will receive Single dose of BAY3389934 as continuous infusion over up to 96 hours.
  Interventions: Drug: BAY3389934
- Dose group 2 of BAY3389934 (Experimental): Subjects will receive Single dose of BAY3389934 as continuous infusion over up to 96 hours.
  Interventions: Drug: BAY3389934
- Dose group 3 of BAY3389934 (Experimental): Subjects will receive Single dose of BAY3389934 as continuous infusion over up to 96 hours.
  Interventions: Drug: BAY3389934
- Dose group 4 of BAY3389934 (Experimental): Subjects will receive Single dose of BAY3389934 as continuous infusion over up to 96 hours.
  Interventions: Drug: BAY3389934

INTERVENTIONS:
Drug: BAY3389934 — Solution for IV infusion

SUMMARY:
Researchers are looking for a better way to treat people who have sepsis induced coagulopathy.

Sepsis happens when bacteria and their toxins spread in the blood, causing an infection. To overcome the infection the body responds activating the immune system, sometimes this immune response is too active and causes uncontrolled blood clot formation, also called sepsis-induced coagulopathy. Sepsis coagulopathy damages blood vessels and organs and leads to low platelet levels in the body. In severe cases, it can even lead to death.

The main purpose of this first in patient study is to learn about how safe BAY 3389934 is, its suitable dose, and how it affects the participants with sepsis induced coagulopathy. For this study, researchers will enroll people receiving treatment for sepsis induced coagulopathy in a hospital intensive care unit (ICU).

For this, the researchers will collect the number of participants with medical problems during and after receiving BAY 3389934. These medical problems are also known as "adverse events". Doctors keep track of all medical problems that happen in studies, even if they do not think they might be related to the study treatments.

Participants will be equally divided into different groups. The first group will receive the lowest dose of BAY 3389934. If researchers consider this dose to be safe, the next group of participants will receive a higher dose until the researchers find a suitable dose of BAY 3389934.

Each participant will be in the study for around 28 days. During the study, the doctors and their study team will:

* Take blood and urine samples,
* Do physical examinations,
* Check vital signs such as body temperature, blood pressure and heart rate,
* Examine heart health using electrocardiogram (ECG)

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥ 18 years of age at the time of signing the informed consent.
* Participants with diagnosed sepsis according to sepsis-3 criteria. Sepsis is defined as life-threatening organ dysfunction caused by a dysregulated host response to infection.
* participants with suspected or documented origin of infection.
* Participants with coagulopathy defined by at least one of the following within 24 hours prior start of study intervention: INR ≥1.40, platelet count in the range of ≥ 30,000/mm3 to < 150,000/mm3 OR greater than 30% decrease in platelets in 24 hours without other known etiology. The platelet count after decrease should not be < 30,000/mm3.
* Participants must be receiving treatment in an ICU.
* Informed consent of capable participant or, in case of participant being incapable of giving informed consent, consent for study inclusion will be sought according to applicable laws and regulations.

Exclusion Criteria:

* Clinically significant active bleeding; known bleeding disorder, history of major traumatic or non-traumatic bleeding (intracranial, retroperitoneal, intraocular) or clinically significant gastrointestinal bleeding within last 6 months.
* Low platelets level or abnormal coagulation status due to any other reason than sepsis.
* Participants with indication for therapeutic dose of: anticoagulation (heparin, argatroban, vitamin K antagonists/warfarin, dabigatran, apixaban, rivaroxaban, edoxaban), oral antiplatelet agents (clopidogrel, ticagrelor, ticlopidine, prasugrel) except low dose (≤100mg) acetyl salicylic acid (ASA), digoxin
* Active malignancy
* Pregnancy or breastfeeding.
* Chronic liver disease Child-Pugh Class C.
* Participants experienced major surgery or major trauma (intrathoracic, intra-abdominal, pelvic or femur) or surgery/trauma in any other area with potentially clinically significant consequences due to bleeding within 28 days before study drug administration.
* Participants experienced neurotrauma or neurosurgery (brain, spine) or orthopedic surgery in spine within 6 months before study drug administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2026-03-16 (Estimated); Study Completion 2026-05-10 (Estimated)

PRIMARY OUTCOMES:
The number of participants with TEAEs (treatment-emergent adverse events) | After the first administration of study intervention to 1 hour after stop from study intervention, up to 97 hours
Severity of TEAEs | After the first administration of study intervention to 1 hour after stop from study intervention, up to 97 hours

SECONDARY OUTCOMES:
Activated partial thromboplastin time (aPTT) | From the first administration of study intervention day 1 to day 6
Prothrombin time (PT) | From the first administration of study intervention day 1 to day 6

CONTACTS AND LOCATIONS:
Locations (20):
- Belgium (4):
  - UZ Antwerpen - Intensive Care, Edegem
  - Centre Hospitalier Universitaire (CHU) de Liege - Domaine Universitaire du Sart Tilman - Intensive Care, Liège
  - Clinique Saint-Pierre d'Ottignies - Intensive Care, Ottignies-Louvain-la-Neuve
  - Universite Catholique de Louvain (UCL) - Cliniques Universitaires Saint-Luc - Intensive Care, Woluwe-Saint-Lambert
- France (7):
  - Centre Hospitalier Universitaire d'Angers - Médecine Intensive Réanimation et Médecine Hyperbare, Angers
  - Hôpital Raymond-Poincaré - Service de Médecine Intensive - Réanimation, Médecine Hyperbare, Garches
  - Centre Hospitalier Départemental Vendée - Service de réanimation polyvalente, La Roche-sur-Yon
  - Centre Hospitalier Universitaire de Limoges Dupuytren 1 - Service de réanimation polyvalente, Limoges
  - Hopital Hotel Dieu Nantes - Service de Médecine Intensive Réanimation, Nantes
  - Hopitaux Universitaires de Strasbourg Nouvel Hopital Civil - Service de Médecine Intensive Réanimation, Strasbourg
  - CHRU de Tours - Hôpital Bretonneau - Médecine Intensive Réanimation, Tours
- Germany (4):
  - Kliniken der Stadt Köln gGmbH - Krankenhaus Merheim - Lungenklinik, Cologne, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus an der Technischen Universitaet Dresden | Medizinische Klinik I - FB Haemostaseologie, Dresden
  - Universitätsklinikum Leipzig AöR | Interdisziplinare Internistische Intensivmedizin, Leipzig
  - Klinikum der Universität München AöR - Klinik für Anaesthesiologie (Campus Großhadern), München
- Netherlands (5):
  - Jeroen Bosch Ziekenhuis - Intensive Care, 's-Hertogenbosch
  - Medisch Spectrum Twente - Intensive Care, Enschede
  - Universitair Medisch Centrum St. Radboud - Intensive Care, Nijmegen
  - Canisius WIlhelmina Ziekenhuis - Intensive Care, Nijmegen
  - Erasmus Medisch Centrum - Intensive Care, Rotterdam

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.